CLINICAL TRIAL: NCT01481649
Title: Risk of Hepatitis B Reactivation After Hematopoietic Stem Cell Transplantation in Donors and Recipients With Prior HBV Exposure
Brief Title: Risk of Hepatitis B Reactivation After Bone Marrow Transplantation With Prior Hepatitis B Virus (HBV) Exposure
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: HKCTR-1422; HKCTR-1422 (Registry Identifier: HKU CTC)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Exposure to Hepatitis B Virus
Keywords: hepatitis B; anti-HBc; HBsAg; HSCT; recipients
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma for hepatitis B virus genotypic, virologic and serologic testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HBsAg-negative, anti-HBc-positive: HBsAg-negative, anti-HBc-positive subjects undergoing hematopoietic stem cell transplantation (HSCT)

SUMMARY:
The purpose of this study is to determine whether preemptive nucleoside analogue therapy or regular virologic monitoring is the preferred method in management patients with prior exposure to hepatitis B vius (HBV) and undergoing hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Occult hepatitis B virus (HBV) reactivation has been documented in bone marrow transplantation recipients who are hepatitis B surface antigen (HBsAg)-negative but with serologic evidence of prior exposure to HBV. However detailed prospective studies documenting the incidence of reactivation and the virologic and serologic kinetics of reactivation are lacking. The investigators prospective study proposes to follow-up 50 such bone marrow transplant recipients with all serologic and virologic parameters monitored every 4 weeks. Patients with detectable HBV DNA will be started on nucleoside analogue therapy. The optimal method and duration of monitoring will also be determined from our study.

ELIGIBILITY:
Inclusion Criteria:

* Documented HBsAg-negative HSCT recipient with or without antibody to the hepatitis B surface antigen (anti-HBs).
* Documented anti-HBc (total)-positive.

Exclusion Criteria:

* Concomitant liver diseases including chronic hepatitis C and D infection, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis.
* Significant alcohol intake (>30 grams per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for hematopoietic stem cell transplantation (HSCT) in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
HBV reactivation (defined as detectable HBV DNA >20 IU/mL) | 2 years
  From date of hematopoietic stem cell transplantation (HSCT) to 2 years after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Kay Seto, MRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Seto WK, Chan TS, Hwang YY, Wong DK, Fung J, Liu KS, Gill H, Lam YF, Lau EHY, Cheung KS, Lie AKW, Lai CL, Kwong YL, Yuen MF. Hepatitis B reactivation in occult viral carriers undergoing hematopoietic stem cell transplantation: A prospective study. Hepatology. 2017 May;65(5):1451-1461. doi: 10.1002/hep.29022. Epub 2017 Mar 22. PMID 28027590